CLINICAL TRIAL: NCT03803748
Title: A Prospective Multicenter, Comparative, Randomized, Double-blind, Non-inferiority Study of Eyestil® Plus Multidose Versus Vismed Multi® in Patients With Moderate to Severe Dry Eye Syndrome
Brief Title: A Non-inferiority Study of Eyestil® Plus Multidose Versus Vismed Multi®
Acronym: 047/SI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 047/SI
Record Dates: First submitted 2018-12-19; First posted 2019-01-15 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-05

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: This is a national, prospective, multicenter, comparative, randomized, double-blinded non-inferiority study performed in two parallel groups.
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eyestil Plus® (Experimental): It's a clinical comparative performance study. Eyestil Plus® eyedrops multidose to be not inferior to Vismed multidose eye drops. Eyestil Plus is an ophthalmic aqueous formulation, multidose sterile preservative free, medical device, class IIB and CE marked. It contains 0.4% sodium hyaluronate. It is not available yet in the French Market.
  The dosage per medical device will be 6 drops a day per dry eye during the three months study period,
  Interventions: Device: Eyestil Plus®
- Vismed (No Intervention): Vismed Multi® is also a sterile multidose preservative free, medical device class IIb and CE marked. It contains 0.18% sodium hyaluronate.
  The dosage per medical device will be 6 drops a day per dry eye during the three months study period.
  The choice of Vismed Multi® as the comparator has been done since it is the current French standard of care treatment for patients with moderate to severe dry eyes.

INTERVENTIONS:
Device: Eyestil Plus® — • To demonstrate the non-inferiority of Eyestil Plus® compared to Vismed Multi® in terms of clinical performance as detected by a reduction of keratitis lesions objectified by staining tests after 1 month of treatment, in patients with moderate to severe dry eye syndrome with keratoconjunctivitis
  Arms: Eyestil Plus®

SUMMARY:
SIFI SpA had developed Eyestil Plus®. It is sterile eyedrops without preservatives with a physiological pH containing sodium hyaluronate. Its intended purpose is to moisturize, lubricate and protect the ocular surface and gives temporary relief to burning, irritation and dry eye-related discomfort, and other complaints induced, for example, by: prolonged use of either soft, semi rigid or rigid contact lenses; exposure to environmental factors (air conditioning, exposure to solar radiation, wind, smoke, pollution, severe climatic conditions, dust); ocular fatigue caused by studying, working, driving or prolonged exposure to electronic devices.

Eyestil Plus® is CE marked but not available yet in all European countries. Considering the European regulatory change on medical devices - from a Directive (Directive 1993/42/EEC) to a Regulation (MDR 2017/745) that now requires clinical evidence of device performance and safety; SIFI Spa decided to implement the present clinical comparative performance study. The choice of Vismed Multi® as the comparator has been done since it is the current French standard of care treatment for patients with moderate to severe dry eyes.

DETAILED DESCRIPTION:
The aim of the study is to demonstrate the non-inferiority of Eyestil Plus® compared to Vismed Multi® in terms of clinical performance as detected by a reduction of keratitis lesions objectified by staining tests after 1 month of treatment, in patients with moderate to severe dry eye syndrome with keratoconjunctivitis. Secondly, the study is aimed at evaluating the safety profile of the product and the patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, male or female, of at least 18 years of age at the screening visit
* Patients understanding the study, willing to follow the instructions and providing their written Informed Consent Form to participate
* Patients with moderate up severe dry eye with keratoconjunctivitis sicca diagnosed at least 4 weeks before the screening visit
* Patients using artificial tears at least once a day for at least 4 weeks months before the screening visit*
* Patients with corneal/conjunctival lesions consistent with a diagnosis of keratoconjunctivitis measured by tests of staining: i.e. the overall score of the corneal staining test must be ≥ 3 and ≤ 9 on the 15-point Oxford scale
* And at least one of the following element:

Tear volume decreased: must be either present a Schirmer test ≥ 3 mm and ≤ 9 mm / 5 minutes or the sum of 3 consecutive measurements of the tear film break-up time (TBUT) ≤ 30s for at least one eye An OSDI score ≥18

- Covered by healthcare insurance.

Exclusion Criteria:

* Patients with medical history of herpetic keratitis, peripheral ulcerative keratitis, sclerites, diabetic retinopathy
* Any systemic disease that is not well controlled for at least 2 months (e.g. lupus, rheumatoid arthritis, thyroiditis…) according to clinical judgment
* Patients using any topical therapies such as non-steroidal anti-inflammatory drugs, cortisone, cyclosporine, vasoconstrictor
* Patients with at least one of the following concomitant ocular inflammatory disease: Stevens Johnson Disease, Atopic Keratoconjunctivitis; Scarlet Eye Pemphigoid
* Patients with anomalies of the eyelid, sucking, infectious conjunctivitis, pterygia, and/or a glaucoma treated with eyedrops
* Presence of graft versus host disease (GVHD)
* Patients who have undergone surgery in the eye, within three months before the study enrolment
* Patients who have undergone corneal transplantation or refractive surgery or plan to undergo any eye surgery in the next four months
* Patients with known or suspected eye allergy
* Patients with a condition or history that, in the opinion of the investigator, may interfere significantly with the subject's participation in the study
* Female pregnant, planning a pregnancy during the study period and nursing an infant
* Patients who are participating or have participated in other clinical trial with investigational drug or device within 30 days prior to screening
* Patients unable to be compliant with the study procedures and requirements, according to the opinion of the investigator
* Patient deprived of liberty by a judicial or administrative decision, or who is under a measure of legal protection (e.g. guardianship or curatorship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Primary endpoint/clinical performance by Oxford scale | between Day 1 and Day 35 ±4
  the between-group comparison of the average variation of the global fluorescein corneal and lissamine green conjunctival staining using the Oxford scale (0 to 15). This refers to the average variation between both timepoints of the Global Ocular Staining Score of the study eye (GOSS) and the comparison between both treatment groups. 0-5 cornea; 0-5 temporal conjuctiva; 0-5 nasal conjunctiva. Max total score: 15

SECONDARY OUTCOMES:
secondary endpoint/clinical performance by TBUT test | between Day 1 and Day 35 ±4 and Day 1 and Day 84 ±7
  The between-group comparisons of the average variation of the time obtained at the TBUT test. This full procedure will be performed 3 times per eye and per time point. At screening and at baseline visits, the sum of these 3 times for at least one eye to be eligible must be ≤ 30 seconds.
  Conventionally TBUT's measures shorter than 10 seconds can be referred to tear film instability and measures shorter than 5 seconds, usually, are undoubtable sign of dry eye. The longer it takes, the more stable the tear film. A short TBUT is a sign of poor tear film. A positive number change from baseline indicates an increase in TBUT (improvement) and a negative number change from baseline indicates a decrease in TBUT (worsening).
secondary endpoint/clinical performance by Oxford scale | between Day 1 and Day 84 ±7 days
  The between-group comparison of the average variation of the global fluorescein corneal and lissamine green conjunctival staining using the Oxford scale. This refers to the average variation between both time points of the Global Ocular Staining Score of the study eye (GOSS) and the comparison between both treatment groups. 0-5 cornea; 0-5 temporal conjuctiva; 0-5 nasal conjunctiva. Max total score: 15
secondary endpoint/clinical performance by Schirmer Test | test between Day 1 and Day 84 ±7
  The between-group comparisons of the average variation of the paper length obtained at the Schirmer test. The Schirmer test without anesthesia will be here performed to measure the rate of secretion of tears produced by the study eye over 5 minutes.The cut-off value for a severe dry eye in the first one is 6 mm. But the cut-off that will here use will be 9 mm with the following interpretation:
  * Normal = ≥ 10 millimeters (mm) of tears,
  * Dry Eye = ≤ 9 mm of tears A positive number change from baseline indicates an increase in tears (improvement) and a negative number change from baseline indicates a decrease in tears (worsening).
secondary endpoint/patient symptoms by Ocular Symptoms Disease Index (OSDI) score | Day 1 and Day 35 ±4 and Day 1 and Day 84 ±7
  The between-group comparisons of the average variation of Ocular Symptoms Disease Index (OSDI) score. The patient's dry eye symptoms will be assessed with the Ocular Surface Disease Index (OSDI). It is a validated 12-questions scale for patients that covers a broad spectrum of ocular surface symptoms, the severity of such symptoms for patients and how these symptoms affect/impact visual function over a 1-week recall period. Its scores range from 0 to 100, with higher scores indicating greater severity of disease.Positive result is considered when the OSDI score is ≥ 18.To be consistent with the IMD indication, patient with moderate to severe dry eye thus with an OSDI ≥ 18 will be selected. If the patient's OSDI score will be strictly below 18 at the screening or baseline visit, s/he will be considered as a screening failure.
secondary endpoint/patient symptoms by Dry Eye-Related Quality -of-Life(DEQS) questionnaire | Day 1 and Day 35 ±4 and [Day 1 and Day 84 ±7
  The between-group comparisons of the average variation of Dry Eye-Related Quality-of-Life (DEQS) questionnaire. It is a validated 15-item scale divided into 2 subscales related to dry eye symptoms and its influence on daily life:
  The frequency is scored on a 5-point Likert scale ranging from 0 (no symptom) to 4 (highest frequency).
  • The degree is scored on a 4-point Likert scale ranging from 1 to 4, a larger number indicates a greater burden.
  The summary score ranges from 0 to 100, higher score indicates higher disability
secondary endpoint/safety | Day 1 and Day 84 ±7
  The description of all adverse events, related and unrelated to the medical devices, anticipated or unanticipated.
secondary endpoint/Investigator overall treatment satisfaction using by a four-point scale | Day 35±4 and Day 84 ±7
  The between group comparison using on a four-point scale assessing investigator's overall satisfaction on the treatment's clinical performance. The between group comparison using on a four-point scale assessing investigator's overall satisfaction on the treatment's clinical performance. Overall investigator' satisfaction of the product's clinical performance will be assessed at the end of the patient follow-up period on a four-point scale from 0: very satisfactory, 1: satisfactory; 2: somewhat unsatisfactory; 3: unsatisfactory Safety • The description of all adverse events, related and unrelated to the medical devices, anticipated or unanticipated.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Jean Pisella, MD, Pr, Principal Investigator — HOPITAL BRETONNEAU
Locations (12):
- France (9):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Chu Morvan, Brest
  - CHU François Mitterand, Dijon
  - Hôpital de la Croix Rousse, Lyon
  - Centre Monticelli, Marseille
  - Hopital La Timone Adultes, Marseille
  - CHU de Nice - Hôpital Pasteur, Nice
  - CHU Saint Etienne/Hôpital Nord, Saint-Etienne
  - Hopital Bretonneau, Tours
- Spain (3):
  - Instituto Oftalmologico Fernandez-Vega, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Recoletas Campo Grande, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided